CLINICAL TRIAL: NCT04735536
Title: A Pilot Electroencephalography (EEG) Study to Evaluate the Effect of CT1812 Treatment on Synaptic Activity in Subjects With Mild to Moderate Alzheimer's Disease
Brief Title: Pilot Clinical Study of CT1812 in Mild to Moderate Alzheimer's Disease Using EEG
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cognition Therapeutics (Industry)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COG0202; RF1AG058710 (NIH); 2019-003552-36 (EudraCT Number)
Record Dates: First submitted 2020-01-30; First posted 2021-02-03 (Actual); Results first posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Single-site, randomized, double-blind, placebo-controlled, 29-day, 2-period crossover Phase 2 study of 1 dose level of CT1812 (active) or placebo in adults with mild to moderate AD.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active Treatment- CT1812 (Experimental): Active Treatment- CT1812 at a dose of 300mg
  Interventions: Drug: CT1812; Other: Placebo
- Control - Placebo (Placebo Comparator): Drug: Placebo Non-active study drug
  Interventions: Drug: CT1812; Other: Placebo

INTERVENTIONS:
Drug: CT1812 — Active Treatment- CT1812 at a dose of 300mg
Other: Placebo — Placebo Comparator

SUMMARY:
This is a single-site, randomized, double-blind, placebo-controlled, 29-day, 2-period crossover Phase 2 study of 1 dose level of CT1812 (active) or placebo in adults with mild to moderate AD.

DETAILED DESCRIPTION:
This is a single-site, randomized, double-blind, placebo-controlled, 29-day, 2-period crossover Phase 2 study of 1 dose level of CT1812 (active) or placebo in adults with mild to moderate AD.

16 participants (8 randomized to 300 mg CT1812, 8 randomly assigned to placebo during each treatment period): the 8 participants randomly assigned to CT1812 in Treatment Period 1 will receive placebo in Treatment Period 2; the 8 participants randomly assigned to placebo in Treatment Period 1 will receive CT1812 in Treatment Period 2.

ELIGIBILITY:
Inclusion Criteria:

1. Women of non-childbearing potential and men, aged 50 to 85 years, inclusive, with a diagnosis of mild to moderate Alzheimer's disease according to the 2018 NIA-AA criteria and at least a 6-month history of decline in cognitive function documented in the medical record.

   i) Non-childbearing potential for women is defined as postmenopausal (last menses greater than 24 months) or undergone a documented bilateral tubal ligation or hysterectomy. If last menses less than 24 months, a serum follicle stimulating hormone (FSH) value confirming post-menopausal status may be used.

   ii) Male participants who are sexually active with a woman of child-bearing potential must agree to use condoms during the study and for 3 months after last dose. Female partners should also consider using an acceptable means of birth control, though it is not mandatory. Acceptable forms of birth control include abstinence, birth control pills, or any double combination of: intrauterine device (IUD), male or female condom, diaphragm, sponge, and cervical cap.
2. CSF positive for amyloid beta (as defined in the study manual). Historical CSF results will be considered provided the results are consistent with the CSF amyloid beta threshold required for inclusion and following discussion with the medical monitor; however, an LP is still required as part of screening procedures
3. Neuroimaging (MRI) consistent with the clinical diagnosis of Alzheimer's disease and without findings of significant exclusionary abnormalities (see Section 9.3 exclusion criteria no. 4). An historical MRI, up to 1 year prior to screening, may be used as long as there have been no interval clinical neurologic events that may suggest a change in the MRI scan.
4. MMSE 18-26 inclusive.
5. Geriatric Depression Scale (GDS) ≤ 6 with no active depression (see Section 9.3 exclusion criteria no. 6).
6. Formal education of 8 or more years.
7. Participants must have a caregiver/study partner who in the opinion of the site's Principal Investigator, has contact with the study participant for a sufficient number of hours per week to provide informative responses on the protocol assessments, oversee the administration of study drug, and is willing and able to participate in all study site visits and some study assessments. The caregiver/ study partner must provide written informed consent to participate in the study.
8. Participants living at home or in the community (assisted living acceptable).
9. Participants must have no known history of difficulty swallowing capsules.
10. Stable pharmacological treatment of any other chronic conditions for at least 30 days prior to screening.
11. Must consent to apolipoprotein E (APOE) genotyping.
12. Participants shall be generally healthy with mobility (ambulatory or ambulatory-aided, ie, walker or cane), vision and hearing (hearing aid permissible) sufficient for compliance with testing procedures.
13. Must be able to complete all screening evaluations.

Exclusion Criteria:

1. Hospitalization (except for planned procedures) or change of chronic concomitant medication within 1 month prior to screening.
2. Participants living in a continuous care nursing facility.
3. Contraindications to the MRI examination for any reason.
4. Screening MRI (or historical MRI, if applicable) of the brain indicative of significant abnormality, including, but not limited to, prior hemorrhage or infarct > 1 cm3, > 3 lacunar infarcts, cerebral contusion, encephalomalacia, aneurysm, vascular malformation, subdural hematoma, hydrocephalus, space-occupying lesion (eg, abscess or brain tumor such as meningioma).
5. Clinical or laboratory findings consistent with:

   1. Other primary degenerative dementia, (dementia with Lewy bodies, fronto-temporal dementia, Huntington's disease, Creutzfeldt-Jakob Disease, Down syndrome, etc).
   2. Other neurodegenerative condition (Parkinson's disease, amyotrophic lateral sclerosis, etc).
   3. Seizure disorder.
   4. Other infectious, metabolic or systemic diseases affecting the central nervous system (syphilis, present hypothyroidism, present vitamin B12 or folate deficiency, other laboratory values etc).
6. A current DSM-V diagnosis of active major depression, schizophrenia or bipolar disorder. Participants with depressive symptoms successfully managed by a stable dose of an antidepressant are allowed entry.
7. Clinically significant, advanced or unstable disease that may interfere with outcome evaluations, such as:

   1. Chronic liver disease, liver function test abnormalities or other signs of hepatic insufficiency (ALT, AST, alkaline phosphatase > 1.5 ULN, lactate dehydrogenase (LDH) > 1.5 x ULN).
   2. Respiratory insufficiency.
   3. Renal insufficiency eGFR < 50 mL/min based on the CKD-EPI formula,
   4. Heart disease (myocardial infarction, unstable angina, heart failure, cardiomyopathy within 6 months before screening).
   5. Bradycardia (< 50/min.) or tachycardia (> 100/min.).
   6. Poorly managed hypertension (systolic > 160 mm Hg and/or diastolic > 95 mm Hg) or hypotension (systolic < 90 mm Hg and/or diastolic < 60 mm Hg).
   7. Uncontrolled diabetes in known diabetics, as defined by hemoglobin A1c (HbA1c) > 7.5.
8. History of cancer within 3 years of screening with the exception of fully excised non-melanoma skin cancers or non-metastatic prostate cancer that has been stable for at least 6 months.
9. Seropositive for human immunodeficiency virus (HIV).
10. History of acute/chronic hepatitis B or C and/or carriers of hepatitis B (seropositive for hepatitis B surface antigen [HbsAg] or anti-hepatitis C [HCV] antibody).
11. Clinically significant abnormalities in screening laboratory tests, including:

    a) Hematocrit less than 35% for males and less than 32% for females, absolute neutrophil cell count of <1500/uL (with the exception of a documented history of a chronic benign neutropenia), or platelet cell count of < 120,000/uL; international normalized ratio (INR) > 1.4 or other coagulopathy, confirmed by repeat assessment.
12. Disability that may prevent the participant from completing all study requirements (e.g., blindness, deafness, severe language difficulty, etc).
13. Within 4 weeks of screening visit or during the study, concurrent treatment with antipsychotic agents, antiepileptics, centrally active anti-hypertensive drugs (e.g., clonidine, l-methyl dopa, guanidine, guanfacine, etc), sedatives, opioids, mood stabilizers (e.g., valproate, lithium); or benzodiazepines, with the following exception:

    a) Low dose lorazepam may be used for sedation prior to MRI scan for those participants requiring sedation. At the discretion of the Investigator, 0.5 to 1 mg may be given orally prior to scan with a single repeat dose given if the first dose is ineffective. No more than a total of 2 mg lorazepam may be used for the MRI scan.
14. Any disorder that could interfere with the absorption, distribution, metabolism or excretion of drugs (eg, small bowel disease, Crohn's disease, celiac disease, or liver disease).
15. Nootropic drugs except stable AD meds (acetylcholinesterase inhibitors and memantine).
16. Suspected or known drug or alcohol abuse, ie, more than approximately 60 g alcohol (approximately 1 liter of beer or 0.5 liter of wine) per day.
17. Suspected or known allergy to any components of the study treatments.
18. Enrollment in another investigational study or intake of investigational drug within the previous 30 days or 5 half-lives of the investigational drug, whichever is longer.
19. Intake of drugs or substances potentially involved in clinically significant induction or inhibition of CYP3A4 or P-gp mediated drug interactions with CT1812, within 4 weeks or 5 half-lives of the interacting drug prior to administration of CT1812 and throughout the study. Grapefruit juice should be avoided in the 2 weeks prior to dosing and throughout the study. See Appendix A for a complete list of prohibited substances.
20. Exposure to immunomodulators, anti Aβ vaccines, passive immunotherapies for AD (e.g., monoclonal antibodies) within the past 180 days and/or exposure to BACE inhibitors within the past 30 days
21. Anticipated use of nonsteroidal anti-inflammatory drugs (NSAIDs) on more than 14 days from Baseline/Day 1 to Day 182. Contraindication to undergoing an LP including, but not limited to: inability to tolerate an appropriately flexed position for the time necessary to perform an LP; international normalized ratio (INR) > 1.4 or other coagulopathy; platelet count of < 120,000/μL; infection at the desired LP site; taking anti-coagulant medication within 90 days of screening (low-dose aspirin is permitted); degenerative arthritis of the lumbar spine; suspected non-communicating hydrocephalus or intracranial mass; prior history of spinal mass or trauma.
22. Any condition, which in the opinion of the Investigator or the Sponsor, makes the participant unsuitable for inclusion.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Everard Vijverberg, MD, Principal Investigator — Brain Research Center, Amsterdam
Locations (1):
- Brain Research Center, Amsterdam, Netherlands

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at a single site in the Netherlands.
Pre-assignment Details: This was a single-site, randomized, double-blind, placebo-controlled, 2 period, crossover, Phase 2 study.
  Eligible participants were randomly assigned to receive either 300 mg/day CT1812 in Period 1 and placebo in Period 2, or placebo in Period 1 and 300 mg/day CT1812 in Period 2 after a washout period of 14 days. The duration of each period was 29 days. A total of 16 participants were randomized and 15 participants completed the study.
Groups:
- First Placebo Non-active Study Drug, Then Active Treatment With CT1812 at a Dose of 300mg; First Active Treatment With CT1812 at a Dose of 300mg, Then Placebo Non-active Study Drug: CT1812 was provided to participants as two hydroxypropyl methylcellulose (HPMC) capsules each containing 150 mg of CT1812. Matching placebo capsules containing lactose monohydrate were provided. CT1812 or matching placebo capsules were to be administered orally as a single daily dose for 29 days. Each dose CT1812 or matching placebo consisted of 2 capsules. All participants ingested the first dose at the study site and were observed for 2 hours. Capsules were swallowed with approximately 240 mL of water with or without food.
Period: Period 1
Arm/Group | First Placebo Non-active Study Drug, Then Active Treatment With CT1812 at a Dose of 300mg | First Active Treatment With CT1812 at a Dose of 300mg, Then Placebo Non-active Study Drug
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Period 2
Arm/Group | First Placebo Non-active Study Drug, Then Active Treatment With CT1812 at a Dose of 300mg | First Active Treatment With CT1812 at a Dose of 300mg, Then Placebo Non-active Study Drug
Started | 8 | 7 (Fifteen participants completed Period 2. Participant 3001-0031 (CT1812/placebo) withdrew consent before Period 2.)
Completed | 8 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo/CT1812: Placebo Non-active study drug/Active Treatment- CT1812 at a dose of 300mg
- CT1812/Placebo: Active Treatment- CT1812 at a dose of 300mg/Placebo: Placebo Comparator
- Total: Total of all reporting groups
Arm/Group | Placebo/CT1812 | CT1812/Placebo | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.6 (6.19) | 67.3 (9.69) | 66.4 (7.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 4 | 4 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 8 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  White | 8 | 8 | 16
  Other | 0 | 0 | 0
Height at Screening [Mean (Standard Deviation); unit: cm] | 175.8 (8.10) | 173.3 (12.34) | 174.5 (10.17)
Body Mass Index at Screening [Mean (Standard Deviation); unit: kg/m^2] | 26.098 (5.4119) | 25.723 (2.6552) | 25.910 (4.1226)
Weight at Screening [Mean (Standard Deviation); unit: Kg] | 81.39 (22.500) | 77.08 (10.021) | 79.23 (16.973)

OUTCOME MEASURES:

1. Primary Outcome: Number of TEAEs, Related TEAEs, SAEs, and Related SAEs
Description: Adverse events were captured from the start of study-related procedures at Visit 1 (including diagnostic assessments or signing of ICF) onward during the course of this study. Adverse events were coded using MedDRA Version 22.0
Time Frame: Up to 126 days
Population: A total of 16 participants were randomized and completed Period 1. Fifteen participants completed Period 2. Participant 3001-0031 (CT1812/placebo) withdrew consent before Period 2. A total of 15 participants completed the study as planned.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Non-active study drug
Arm/Group | Placebo | CT1812
Number analyzed (Participants) | 15 | 16
Participants
  All TEAEs | 6 | 11
  Mild TEAEs | 4 | 7
  Moderate TEAEs | 2 | 4
  Severe TEAEs | 0 | 0
  Related TEAEs | 3 | 3
  TEAEs Leading to Treatment Discontinuation | 0 | 0
  SAEs | 0 | 0
  Related SAEs | 0 | 0

2. Primary Outcome: Change in the Brain Activity Reflected by Changes of Spectral Power in Conventional Frequency Bands Measured by the Global Relative Theta (4-8 Hz) Power Obtained Through EEG Assessment.
Description: Global relative theta power was quantified and summarized descriptively (observed values, change from the pre-treatment values) by treatment and time point using the Safety Population. The change from period baseline in global relative theta power within each period was analyzed using a linear mixed model with fixed effects for treatment group (CT1812 or placebo), sequence, and period, and a random effect for subject within sequence. The analysis was conducted using PROC MIXED. The ability of CT1812 to rapidly restore synapse number to normal was expected to result in a decrease in EEG theta power in AD patients in response to short-term treatment with CT1812. Thus, a decrease in the Global Relative Theta Power represents better outcomes, while high values in the Global Relative Theta Power represent worse outcomes. The unit is represented by uV^2/Hz (microvolt squared per frequency). This is a common unit for spectral power density, and how relative power measures are displayed.
Time Frame: Day 1 through Day 29 of Period 1 and Day 1 (study day 44) and Day 29 (study day 72) of Period 2
Population: Up to 16 participants were planned to be enrolled. A total of 16 participants were randomized and completed Period 1. Fifteen participants completed Period 2. Participant 3001-0031 (CT1812/placebo) withdrew consent before Period 2. A total of 15 participants completed the study as planned.
Measure: Mean (Standard Deviation); unit: uV^2/Hz
Groups:
- Placebo: Placebo Non-active study drug
- CT1812: Active Treatment- CT1812 at a dose of 300mg/Placebo
Arm/Group | Placebo | CT1812
Number analyzed (Participants) | 15 | 16
uV^2/Hz
  Global Relative Theta Power Day 1 | 0.2133 (0.06158) | 0.2071 (0.08209)
  Global Relative Theta Power Day 29: number analyzed (Participants) | 14 | 16
  Global Relative Theta Power Day 29 | 0.2276 (0.07872) | 0.1971 (0.07569)
  Change from Day 1 to Day 29: number analyzed (Participants) | 14 | 16
  Change from Day 1 to Day 29 | 0.0104 (0.03210) | -0.0100 (0.04280)

3. Primary Outcome: Changes in Predose CT1812 Plasma Concentrations.
Description: For the measurements of pre-dose and post-dose plasma concentrations of CT1812, samples were collected 1± 0.25 hour predose. Single concentrations of CT1812 at selected predose and post-dose time points were reported.
Time Frame: Baseline through Day 84: Pre and Post- Dose on Days 1, 29 AND Pre Dose Days 8, 15, 22.
Population: The pharmacokinetic (PK) population was comprised of all randomized participants who received at least one dose of study drug and had at least one PK concentration of CT1812. All 16 randomized participants were included in the PK Population.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- CT1812: All 16 randomized participants were included in the PK Population.
Arm/Group | CT1812
Number analyzed (Participants) | 16
ng/mL
  Period Day 1, Predose | 0.00 (0.000)
  Period Day 1, Post-dose | 179.64 (136.717)
  Period Day 8, Predose | 25.49 (25.017)
  Period Day 15, Predose | 14.93 (7.826)
  Period Day 22, Predose | 13.76 (8.000)
  Period Day 29, Predose | 14.08 (8.984)
  Period Day 29, Post-dose | 169.20 (246.150)

4. Primary Outcome: Changes in Predose CT1812 Plasma Concentrations.
Description: as for outcome 3
Time Frame: Baseline through Day 84: Pre and Post- Dose on Days 1, 29 AND Pre Dose Days 8, 15, 22.
Population: as for outcome 3
Measure: Median (Full Range); unit: ng/mL
Arm/Group | CT1812
Number analyzed (Participants) | 16
ng/mL
  Period Day 1, Post-dose | 161.50 [4.1 to 406.0]
  Period Day 8, Predose | 23.05 [2.5 to 106.0]
  Period Day 15, Predose | 13.20 [2.9 to 28.6]
  Period Day 22, Predose | 12.40 [3.6 to 28.8]
  Period Day 29, Predose | 12.60 [2.6 to 36.0]
  Period Day 29, Post-dose | 96.35 [7.5 to 949.0]

ADVERSE EVENTS:
Time Frame: 126 days
Arm/Group | Placebo | CT1812
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/16
Other Adverse Events (participants affected / at risk) | 6/15 | 11/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=15) | CT1812 (N=16)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Burns first degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural headache (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Hematoma (Vascular disorders) | 1 (1) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Corona virus infection (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-02-21): https://cdn.clinicaltrials.gov/large-docs/36/NCT04735536/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-20): https://cdn.clinicaltrials.gov/large-docs/36/NCT04735536/SAP_001.pdf